CLINICAL TRIAL: NCT03371992
Title: Pilot Study of the Nilogen Ex-Vivo Assay (3D-EX) and Its Ability to Predict Therapeutic Response to Anti-PD1 (Nivolumab, Embrolizumab) or Anti-PDL1(Atezolizumab) in Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Pilot Study of Nilogen 3D-EX and Its Ability to Predict Therapeutic Response to Anti-PD1 or Anti-PDL1 in NSCLC
Acronym: NO3DEXPL
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nilogen Oncosystems (Industry)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NO88352235
Record Dates: First submitted 2017-12-03; First posted 2017-12-13 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: immunotherapy; anti-PD1; anti-PDL1; biomarker; drug mechanism
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; pembrolizumab; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lung Cancer Patients (Other): Lung cancer patients receiving one of three standard of care immunotherapy drugs including nivolumab, pembrolizumab or atezolizumab. 3D-EX will be performed on biopsies from patients enrolled in the study to correlate with the patient's evaluation of response by RECIST.
  Interventions: Drug: Nivolumab; Diagnostic Test: 3D-EX; Other: Evaluation of Response by RECIST

INTERVENTIONS:
Drug: Nivolumab — Nivolumab, pembrolizumab or atezolizumab will be administered as per the established standard of care for the eligible population.
  Other Names: pembrolizumab; atezolizumab
Diagnostic Test: 3D-EX — Analysis of drug-mediated changes in the tumor microenvironment.
  Other Names: 3D ex vivo assay
Other: Evaluation of Response by RECIST — Evaluation of tumor response using the set of published rules to determine if a tumor has responded, is stable or progressed during treatments.

SUMMARY:
Subjects will be eligible for this study if they are about to start on a drug called nivolumab for lung cancer. Some patients' cancers respond to nivolumab but a majority of patients do not. To better determine which patients will most likely respond to nivolumab or not, the investigators are testing an assay that tests biopsy tissue to determine if the subject's tumor will likely respond to nivolumab.

The main purpose of this research study is to see if this specialized test can help identify people with locally advanced or metastatic non-small cell lung cancer who are more likely to benefit from treatment with nivolumab. The results of the tests will not affect whether or not subjects receive nivolumab but may help identify future patients who are more likely to benefit from nivolumab. The study assay is extra and experimental.

DETAILED DESCRIPTION:
Overview of PD-1 inhibition for locally advanced or metastatic NSCLC Lung cancer (LC) is the most common malignancy-related death in the United States (causing deaths in ~ 86,380 men and ~71,660 women in 2015. Fifteen percent of LC patients present with Stage I disease, which is treated primarily with surgery, leading to a 5-year survival rate of 54%. Approximately 57% of LC patients are initially diagnosed with metastatic disease (Stage IV) with a corresponding 5-year survival rate of 4.2%.

More recently, major treatment responses have been observed with the use of immune checkpoint inhibitor proteins expressed on the surface of lymphocytes and other immune cells, most notably on cytotoxic T-cells. When bound to their specific ligand, often another surface-bound protein on a neighboring cell, they can transmit stimulatory or inhibitory signals to activate or inhibit the cellular adaptive immune response. Several studies showed that the predominant mechanism by which NSCLC evades detection and elimination by the immune system is by exploiting one such inhibitory pathway through the expression of programmed death ligand 1 (PD-L1, B7-H1). PD-L1 then binds to its receptor, programmed cell death protein 1 (PD1), on surveilling lymphocytes and initiates a signaling cascade which leads to lymphocyte exhaustion, a state of impaired function. The most successful immune checkpoint inhibitors so far are anti PD1 or anti-PD-L1 monoclonal antibodies that prevent PD1-PD-L1 interaction at the tumor-immune interface. In this pilot study, the investigators will investigate if Nilogen's functional ex vivo bioassay can predict therapeutic response to anti PD1 (nivolumab, pembrolizumab) or anti PD-L1 (atezolizumab) in advanced non-small cell lung cancer (NSCLC).

Functional bioassay as a potential predictive biomarker. The intent of using anti-PD-1/PD-L1 as an anti-cancer therapeutic is to block one of the ways that tumors inhibit T cell function within the tumor microenvironment, allowing restoration of T cell function. Therefore, the investigators hypothesize that a bioassay that directly measures restoration of T cell function in the context of all of the elements of the tumor microenvironment could accurately predict whether or not a patient will be clinically responsive to a particular immunotherapeutic agent that is designed to target the tumor microenvironment. A tumor biopsy from a patient who will be clinically responsive to anti-PD-1 will contain inactive T cells that may have their functional activity restored by the provision of anti-PD-1/PD-L1 ex vivo, much like what is seen in the ex vivo experiments performed at Nilogen using the 3D-EX platform (www.nilogen.com). To assess tumor response to nivolumab, pembrolizumab or atezolizumab the investigators will use their proprietary immune cell function analysis in tumor samples obtained by FNA biopsy upon treatment with nivolumab, pembrolizumab or atezolizumab, pembrolizumab or atezolizumab ex vivo.

Hypothesis

1. In 80% of patients, FNA samples will provide a sufficient number of viable tumor cells to perform ex vivo functional bioassays with nivolumab, pembrolizumab or atezolizumab.
2. Patients whose tumor FNA samples fail to respond to nivolumab, pembrolizumab or atezolizumab, in the 3D Ex-Vivo assays will likely not show a clinical response to systemic nivolumab, pembrolizumab or atezolizumab treatment.

Study Objectives

Primary Objective To test whether it is feasible to perform the 3D-EX functional response bioassay in the context of patients with advanced NSCLC receiving treatment with nivolumab, pembrolizumab or atezolizumab in a standard clinical setting.

Overall study design Eligible patients will have a histologic or cytologic diagnosis of NSCLC; advanced-stage disease who are appropriate candidates for therapy with nivolumab, pembrolizumab or atezolizumab, and age greater than 18 years. Prior surgery, chemotherapy and/or radiotherapy are allowed. Inclusion and exclusion criteria are outlined in the appropriate section. All inclusion and exclusion criteria will be assessed within 6 weeks prior to the first dose of nivolumab, pembrolizumab or atezolizumab. Baseline radiographic studies should be performed within 30 days of screening. This clinical study will require central IRB approval. Informed consent will be obtained from each patient prior to screening and enrolling in the study.

Nivolumab, pembrolizumab or atezolizumab will be administered as per the established standard of care for the eligible population.

Prediction of Response to Nivolumab, pembrolizumab or atezolizumab by Nilogen's 3D-EX Bioassay.

In previous preclinical and clinical studies the investigators showed that FNA samples provide a sufficient number of viable tumor cells to perform drug sensitivity assays ex-vivo. The assay protocol is optimized to process tumor FNA samples, where the tumor microenvironment is intact and contains tumor cells and all other tumor-infiltrating inflammatory cells as well as specialized tumor stroma. Prior to initiation of therapy, tumor samples will be collected by FNA from accessible tumor tissue. For the ex vivo assays, aspirates will be obtained from each patient after collection of biopsy samples required for SOC. The FNA samples will be immediately shipped to the Nilogen Laboratory. All proposed assays will be performed at the Nilogen Oncosystems laboratory in Tampa, FL according to CLIA standards.

Patients who do not have a site of disease that will provide enough tumor cells for analyses will be taken off study. In adequate samples, tumor FNA samples will be treated nivolumab, pembrolizumab or atezolizumab at clinically relevant concentrations. At the end of incubation T-cell activation will be assessed by a proprietary approach including evaluation of drug-mediated changes in three parameters: (1) T-cell activation, (2) cytokine release and (3) gene expression profiles. The response rate to treatment will be scored for T-cell activity and correlated with patient outcome.

The investigators hypothesize that tumors that fail to respond ex vivo will not be likely to be responsive in vivo in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

1. Be willing and able to provide written informed consent for the trial.
2. Be at least 18 years of age on the day of signing informed consent.
3. Have a histologic or cytologic diagnosis of Stage IV NSCLC.
4. Must be medically eligible to receive nivolumab, pembrolizumab or atezolizumab as the standard of care for the next line of therapy (must have previously received first line platinum doublet chemotherapy) as determined by their oncologist.
5. Have measurable disease based on RECIST 1.1 (see section 7.1 or appropriate number).
6. Be willing and medically fit to undergo a fresh (newly obtained) diagnostic biopsy of a metastatic lesion or primary site of disease before receiving nivolumab, pembrolizumab or atezolizumab. "Fresh (newly-obtained)" is defined as a specimen obtained up to 6 weeks prior to initiation of treatment with nivolumab, pembrolizumab or atezolizumab on Day 1.
7. Fit in either of these categories:

   1. Stage I-III NSCLC patients who develop metastatic disease within 6 months of receiving definitive (curative) treatment that includes platinum-based chemotherapy, and who require biopsy for either confirmation of diagnosis or further molecular or immunohistochemical testing to guide treatment.
   2. Stage IV NSCLC patients with progression of disease following platinum based chemotherapy, and who require biopsy for either confirmation of diagnosis or further molecular or immunohistochemical testing to guide treatment.
   3. Stage IV NSCLC patients who will receive nivolumab, pembrolizumab or atezolizumab as the standard of care in special circumstances (eg, when chemotherapy is contraindicated or if a patient declines to be treated with chemotherapy).
8. Be willing to undergo at least 4 fine needle aspirations for experimental purposes at the time of the standard of care biopsy.
9. Have a performance status of 0 or 1 on the ECOG Performance Scale.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating in and receiving therapy as part of a different clinical trial.
2. Is not a candidate to receive nivolumab, pembrolizumab or atezolizumab as determined by the patient's oncologist.
3. Has an active infection requiring systemic therapy.
4. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might; (1) confound the results of the trial, (2) that would substantially increase risk of incurring adverse events (AEs) from nivolumab, pembrolizumab or atezolizumab, (3) that would interfere with the subject's participation for the full duration of the trial, or (4) is not in the best interest of the subject to participate, in the opinion of the treating investigator.
5. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
6. Is pregnant or breastfeeding.
7. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
8. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-03-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of target lesions by RECIST | Tumor size is assessed via CT every 8 weeks and RECIST criteria will be documented every 8 weeks after the first treatment for progression or date of death, whichever comes first, for up to 60 months.
  Complete Response (CR) is defined as disappearance of all target lesions Partial Response (PR) is defined as at least a 30% decrease in the sum of longest dimension (LD) of target lesions taking as reference the baseline sum LD Progressive Disease (PD) is defined as at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started

CONTACTS AND LOCATIONS:
Overall Officials: Soner Altiok, MD, PhD, Principal Investigator — Nilogen Oncosystems; Igor Rybkin, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health Systems, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared but the results of the clinical trial will be published in a peer-reviewed journal.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Brahmer JR, Pardoll DM. Immune checkpoint inhibitors: making immunotherapy a reality for the treatment of lung cancer. Cancer Immunol Res. 2013 Aug;1(2):85-91. doi: 10.1158/2326-6066.CIR-13-0078. Epub 2013 Jul 22. PMID 24777499
- [Background] Taube JM, Klein A, Brahmer JR, Xu H, Pan X, Kim JH, Chen L, Pardoll DM, Topalian SL, Anders RA. Association of PD-1, PD-1 ligands, and other features of the tumor immune microenvironment with response to anti-PD-1 therapy. Clin Cancer Res. 2014 Oct 1;20(19):5064-74. doi: 10.1158/1078-0432.CCR-13-3271. Epub 2014 Apr 8. PMID 24714771
- [Background] Jiang Y, Li Y, Zhu B. T-cell exhaustion in the tumor microenvironment. Cell Death Dis. 2015 Jun 18;6(6):e1792. doi: 10.1038/cddis.2015.162. PMID 26086965
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, Patnaik A, Aggarwal C, Gubens M, Horn L, Carcereny E, Ahn MJ, Felip E, Lee JS, Hellmann MD, Hamid O, Goldman JW, Soria JC, Dolled-Filhart M, Rutledge RZ, Zhang J, Lunceford JK, Rangwala R, Lubiniecki GM, Roach C, Emancipator K, Gandhi L; KEYNOTE-001 Investigators. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28. doi: 10.1056/NEJMoa1501824. Epub 2015 Apr 19. PMID 25891174
- [Background] Fehrenbacher L, Spira A, Ballinger M, Kowanetz M, Vansteenkiste J, Mazieres J, Park K, Smith D, Artal-Cortes A, Lewanski C, Braiteh F, Waterkamp D, He P, Zou W, Chen DS, Yi J, Sandler A, Rittmeyer A; POPLAR Study Group. Atezolizumab versus docetaxel for patients with previously treated non-small-cell lung cancer (POPLAR): a multicentre, open-label, phase 2 randomised controlled trial. Lancet. 2016 Apr 30;387(10030):1837-46. doi: 10.1016/S0140-6736(16)00587-0. Epub 2016 Mar 10. PMID 26970723
- [Background] Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J, Gadgeel SM, Hida T, Kowalski DM, Dols MC, Cortinovis DL, Leach J, Polikoff J, Barrios C, Kabbinavar F, Frontera OA, De Marinis F, Turna H, Lee JS, Ballinger M, Kowanetz M, He P, Chen DS, Sandler A, Gandara DR; OAK Study Group. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet. 2017 Jan 21;389(10066):255-265. doi: 10.1016/S0140-6736(16)32517-X. Epub 2016 Dec 13. PMID 27979383
- [Background] Butte MJ, Keir ME, Phamduy TB, Sharpe AH, Freeman GJ. Programmed death-1 ligand 1 interacts specifically with the B7-1 costimulatory molecule to inhibit T cell responses. Immunity. 2007 Jul;27(1):111-22. doi: 10.1016/j.immuni.2007.05.016. Epub 2007 Jul 12. PMID 17629517
- [Background] Stamper CC, Zhang Y, Tobin JF, Erbe DV, Ikemizu S, Davis SJ, Stahl ML, Seehra J, Somers WS, Mosyak L. Crystal structure of the B7-1/CTLA-4 complex that inhibits human immune responses. Nature. 2001 Mar 29;410(6828):608-11. doi: 10.1038/35069118. PMID 11279502
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Rubio-Viqueira B, Mezzadra H, Nielsen ME, Jimeno A, Zhang X, Iacobuzio-Donahue C, Maitra A, Hidalgo M, Altiok S. Optimizing the development of targeted agents in pancreatic cancer: tumor fine-needle aspiration biopsy as a platform for novel prospective ex vivo drug sensitivity assays. Mol Cancer Ther. 2007 Feb;6(2):515-23. doi: 10.1158/1535-7163.MCT-06-0388. PMID 17308050
- [Background] Hidalgo M, Amador ML, Jimeno A, Mezzadra H, Patel P, Chan A, Nielsen ME, Maitra A, Altiok S. Assessment of gefitinib- and CI-1040-mediated changes in epidermal growth factor receptor signaling in HuCCT-1 human cholangiocarcinoma by serial fine needle aspiration. Mol Cancer Ther. 2006 Jul;5(7):1895-903. doi: 10.1158/1535-7163.MCT-05-0525. PMID 16891476